CLINICAL TRIAL: NCT00648700
Title: Single-Dose Fasting In Vivo Bioequivalence Study of Levothyroxine Sodium Tablets (300 μg; Mylan) to Levothroid® Tablets (300 μg; Llyod) in Healthy Volunteers.
Brief Title: Fasting Study of Levothyroxine Sodium Tablets 300 μg to Levothroid® Tablets 300 μg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LEVO-0573
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Thyroxine

ARMS (2):
- 1 (Experimental): Levothyroxine Sodium Tablets 300 μg
  Interventions: Drug: Levothyroxine Sodium Tablets 300 μg
- 2 (Active Comparator): Levothroid® Tablets 300 μg
  Interventions: Drug: Levothroid® Tablets 300 μg

INTERVENTIONS:
Drug: Levothyroxine Sodium Tablets 300 μg — 2x300mcg, single dose fasting
  Arms: 1
Drug: Levothroid® Tablets 300 μg — 2x300mcg, single dose fasting
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's levothyroxine sodium 300 μg tablets to Lloyd's Levothroid® 300 μg tablets following a single 600 μg (2 x 300 μg) dose administered in healthy adult volunteers under fasting conditions. Statistical analysis of the data revealed that 90% confidence intervals were within the acceptable bioequivalent range of 80% and 125% for the natural log transformed parameters LNAUC0-48hr and LNCPEAK for baseline corrected total levothyroxine.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-50 years.
2. Sex: Men and/or non-pregnant, non-lactating women.

   1. Women of childbearing potential must have negative serum β human chorionic gonadotropin (HCG) pregnancy tests performed within 14 days prior to of the study and on the evening prior to each dose administration. An additional serum (β HCG) pregnancy test will be performed upon completion of the study.
   2. Women of childbearing potential must practice abstinence or be using an acceptable form of contraception throughout the duration of the study. Oral contraceptives are not to be used within 3 months prior to dosing and throughout the course of the study due to the fact that they increase serum TBG concentrations, and therefore, elevate T4. Acceptable forms of contraception include the following:

      1. intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
      2. barrier methods containing or used in conjunction with a spermicidal agent, or
      3. postmenopausal accompanied with a documented postmenopausal course of at least one year or surgical sterility (tubal ligation, oophorectomy or hysterectomy).
3. Weight: At least 60 kg (132 lbs) for men and 48 kg (106 lbs) for women, and within 15% of Ideal Body Weight (IBW), as referenced by the Table of "Desirable Weights of Adults" Metropolitan Life Insurance Company, 1983 (See Part II Administrative Aspects of Bioequivalence Protocols).
4. All subjects should be judged normal (euthyroid) and healthy during a prestudy medical evaluation (physical examination, laboratory evaluation, blood chemistry, serum T4 (free and total), serum T3 (total only), serum thyroid-stimulating hormone (TSH), serum thyroxine-binding globulin (TBG), hepatitis B and hepatitis C tests, HIV test, 12-lead ECG, and urine drug screen including amphetamine, barbiturates, benzodiazepine, cannabinoid, cocaine, opiate screen, phencyclidine, and methadone) performed within 14 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco-containing products within 1 year of the start of the study.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. A positive test for any drug included in the urine drug screen.
   6. History of drug and/or alcohol abuse.
3. Medications:

   1. Use of any prescription or over-the-counter (OTC) medications within the 30 days prior to the initial dose of study medication. These may include but is not limited to: infant soybean formula, steroids, salicylates, preparations containing iodine, such as vitamins; oral anti-diabetic agents; all resins for lowering of cholesterol, such as cholestyramine; sucralfate, propranolol, amiodarone, phenytoin, carbamazepine, furosemide; aluminum-containing antacids, including aluminum hydroxide; rifampin, calcium channel blockers and ferrous sulfate.
   2. Use of any hormonal contraceptives or hormone replacement therapy within 3 months prior to study medication dosing.
   3. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, or neurologic disease.
   2. Acute illness at the time of either the pre-study medical evaluation or dosing.
   3. A positive HIV, hepatitis B, or hepatitis C test.
   4. History of any thyroid disease.
   5. Subjects with any underlying medical condition known to interfere with the absorption or metabolism of thyroid hormones.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
   3. Any thyroid function test outside normal limits.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Subjects who received any surgical treatment within 6 months prior to the initial dose of study medication.
9. Subjects with known allergies or hypersensitivity to thyroid preparations or their inactive ingredients.
10. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
11. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.
12. Consumption of products containing walnuts, cotton seed meal, soybean flour or dietary fiber within 48 hours of drug administration.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2005-08; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D., Principal Investigator — PRACS Institute Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html